CLINICAL TRIAL: NCT01758757
Title: Comparison of Small-gauge and Conventional Vitrectomy for Proliferative Diabetic Retinopathy
Brief Title: Comparison of Small-gauge Vitrectomy and Conventional Vitrectomy for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Kyorin Eye Center, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Kyorineye010; Vitrectomy for PDR
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-12

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative diabetic retinopathy; Vitrectomy
MeSH Terms: interventions — Vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Proliferative diabetic retinopathy (Active Comparator)
  Interventions: Procedure: Vitrectomy

INTERVENTIONS:
Procedure: Vitrectomy

SUMMARY:
Surgical outcome of vitreous surgery for proliferative diabetic retinopathy (PDR) with conventional 20, 23, and 25-gauge vitrectomy were compared.

DETAILED DESCRIPTION:
The 424 eyes of 347 patients of PDR who underwent vitreous surgery for persistent vitreous hemorrhage or progressive proliferative membrane were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patients of proliferative diabetic retinopathy who underwent vitreous surgery and followed at least 6 months

Exclusion Criteria:

* The patients of proliferative diabetic retinopathy who underwent vitreous surgery but did not follow more than 6 months.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2007-09; Primary Completion 2011-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Incidence of retinal breaks | One year

SECONDARY OUTCOMES:
Incidence of neovascular glaucoma | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Study Chair — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan

REFERENCES:
- [Derived] Yokota R, Inoue M, Itoh Y, Rii T, Hirota K, Hirakata A. Comparison of microinsicion vitrectomy and conventional 20-gauge vitrectomy for severe proliferative diabetic retinopathy. Jpn J Ophthalmol. 2015 Sep;59(5):288-94. doi: 10.1007/s10384-015-0396-y. Epub 2015 Jul 23. PMID 26202442